CLINICAL TRIAL: NCT05730738
Title: Effect of Dalfampridine on Gait Impairment, Cognition and Fatigue in Egyptian Patients With Multiple Sclerosis
Brief Title: Dalfampridine in Egyptian Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ali Shalash, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU MD 551/2020
Record Dates: First submitted 2021-12-05; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis,; Dalfampridine; Gait; cognition; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with MS will be evaluated for inclusion and exclusion criteria using the selected screening scales. Eligible patients will be randomly assigned to one of two groups: dalfampridine ER 10mg twice daily group and placebo group for 12 consecutive weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomization was done by a research randomization, The copy of the randomization table of patients to the 2 groups was kept with 2 different personnel not working on the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dalfampridine (Active Comparator): patients received dalfampridine ER 10mg twice daily
  Interventions: Drug: Dalfampridine ER, 10 Mg Oral Tablet, Extended Release
- Placebo (Placebo Comparator): patients received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine ER, 10 Mg Oral Tablet, Extended Release — The only approved treatment for impaired ambulation in MS is Dalfampridine (also known as fampridine, 4-aminopyridine, 4-AP). Fampridine penetrates the blood-brain barrier and improves impaired axonal conduction by selectively blocking potassium channels
  Arms: dalfampridine
Drug: Placebo — placebo similar to Dalfampridine capsule
  Arms: Placebo

SUMMARY:
The only approved treatment for impaired ambulation in MS is Dalfampridine (also known as fampridine, 4-aminopyridine, 4-AP). Fampridine penetrates the blood-brain barrier and improves impaired axonal conduction by selectively blocking potassium channels. Moreover, further studies investigated the possible beneficial effect of dalfampridine on cognitive functions and fatigue.

The main objective of this study is to investigate the effect of dalfampridine on gait impairment, cognitive functions and fatigue in a sample of Egyptian patients with multiple sclerosis.

DETAILED DESCRIPTION:
Type of the Study: randomized double blinded placebo controlled study. Study Setting: MS outpatient clinic in Ain Shams University hospital and Dar Alshefa Hospital, they are located in Eastern Cairo and serves large sector of the ministry of health patients in Greater Cairo.

Period two years. Population patients with relapsing remittent multiple sclerosis attending to ms clinic meeting the inclusion criteria.

Sample size: 100 patients (50 patients in active group and 50 patients in placebo group).

Study Procedures:

Patients diagnosed with MS will be evaluated for inclusion and exclusion criteria using the selected screening scales. Eligible patients will be randomly assigned to one of two groups: dalfampridine ER 10mg twice daily group and placebo group for 12 consecutive weeks.

All patients will be subjected to:

Comprehensive medical history and neurological examination. Demographic information (sex, age and education years), as well as clinical characteristics of them (age at onset, duration of illness, onset of last relapse, received DMD and other medications during the study).

MRI brain and spine lesions (site & number of lesions). Check list for side effects of dalfampridine. Expanded Disability Status Scale (EDSS) (Kurtzke, 1983). The Patient Health Questionnaire (PHQ-9) Arabic translation (Kroenke et al., 2001).

Gait assessment by:

* Timed 25 foot walk test (25FWT) (Motl et al., 2017).
* Hauser ambulatory index (Hauser et al., 1983).
* Berg balance scale (Berg et al., 1992).
* Falls in last 2 weeks.

Cognitive assessment by:

* Arabic validated version of the BICAM battery, which compromised the symbol digit modality test (SDMT, information processing speed), verbal learning test (VLT, verbal memory) and brief visuospatial memory teat revised (BVMT-R, visual memory) (Alboudi et al., 2020).
* Montreal Cognitive Assessment (MoCA) Arabic version (Abd El-Rahman and El-Gaafary, 2009).
* Frontal assessment battery (FAB) (for executive functions) (Dubois and Litvan, 2000).

Fatigue assessment by:

o Modified fatigue impact scale (MFIS) in last 4 weeks Arabic version (Farran et al., 2020).

• Assessment for gait, cognition and fatigue will be done at baseline and after 12 weeks of treatment by a blinded rater.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Individuals diagnosed with RRMS based on revised McDonald Criteria 2017
* Patients with Expanded Disability Status Scale (EDSS) ≤ 5.5
* Patients with gait impairment according to 25 foot walk test (25FWT) with cutoff ≥ 4 seconds

Exclusion Criteria:

* Women who are pregnant, intended to be pregnant or breastfeeding.
* Past History of epilepsy or trigeminal neuralgia.
* History of any psychiatric or medical illness affecting cognition and fatigue.
* Other comorbidities that might affect gait.
* Clinical relapse in the last three months.
* Uncooperative patients or couldn't perform the required scales.
* Patients with moderate to severe depression according to patient health questionnaire (PHQ-9) with cutoff point ≥15.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
gait | at 3 months
  Timed 25 foot walk test (25FWT), higher scores mean a worse outcome
gait | 3 months
  Hauser ambulatory index, higher scores mean a worse outcome
Balance | 3 months
  Berg balance scale, higher scores mean a worse outcome

SECONDARY OUTCOMES:
cognition | 3 months
  Arabic validated version of the BICAM battery
fatigue | 3 months
  Modified fatigue impact scale: physical, 0 to 36; cognitive, 0 to 40; and psychosocial, 0 to 8. higher scores mean a worse outcome
cognition | 3 months
  MOCA, higher scores mean a better outcome
Cognition | 3 months
  frontal assessment battery

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided